CLINICAL TRIAL: NCT00304564
Title: Fall Prevention and The Nolwenn Effect in Texas Geriatric Nursing Home Settings
Brief Title: Study of the Effect of the Music of Nolwenn Leroy in Fall Prevention Strategies in Texas Nursing Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carrick Institute for Graduate Studies (Other)
Responsible Party: Principal Investigator, Frederick Carrick, PhD, FACCN, Principal Investigator, Carrick Institute for Graduate Studies
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CI-02-01-06-02
Record Dates: First submitted 2006-03-15; First posted 2006-03-20 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Accidental Falls
Keywords: Posturography, Fall Prevention, Geriatrics, Nolwenn Effect

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- geriatric community (Experimental): Subject will stand on a computerized posturography force plate and stability scores are measured
  Interventions: Behavioral: Music Listening

INTERVENTIONS:
Behavioral: Music Listening — subjects listen to music

SUMMARY:
Falls are the largest cause of death in the elderly and those in nursing homes have even a higher incidence of falling. The purpose of this study is to determine whether listening to the Music of Nolwenn Leroy daily is effective in fall prevention in those elderly patients who are residents in several Texas geriatric nursing home facilities. The music of Nolwenn Leroy has been shown to be effective in fall reduction in a different setting (Posturographic Changes and Fall Prevention associated with Music Therapy: The Nolwenn Effect (USA ClinicalTrials.gov Identifier: NCT00121693) )with results better than listening to Mozart of any other music. Another similar study (USA ClinicalTrials.gov Identifier:NCT00272272)is presently being conducted in a geriatric nursing home facility in Georgia. Dynamic posturographic measurments will be obtained from all residents and compared to normative age related data and utilized to measure stability changes in this study.

DETAILED DESCRIPTION:
Falls are a serious health issue and are the greatest cause of death in the elderly. The use of the music of Nolwenn Leroy in fall prevention has been reported at a major scientific meeting "Posturographic Changes and Fall Prevention associated with Music Therapy: The Nolwenn Effect (USA ClinicalTrials.gov Identifier: NCT00121693) featured at the 7th Annual American Music Therapy Association Conference in Orlando, Florida, Nov 15-20, 2005 and Decreasing falls in a geriatric nursing home setting is associated with the saving of lives. Another similar study (USA ClinicalTrials.gov Identifier:NCT00272272)is presently being conducted in a geriatric nursing home facility in Georgia. We propose the utilization of the Nolwenn Effect in our resident geriatric population at several Dallas, Texas Geriatric Nursing Home Facilities and comparing fall rates to those we have carefully recorded in the past. We will obtain computerized dynamic posturographic measurements utilizing the CAPS posturographic unit by Vestibular Technologies on all residents of several Dallas Geriatric Nursing Facilities. Our findings will be compared to normative data previously validated to represent a probability of falling. Daily listening to selections from Nolwenn Leroy's CD "Nolwenn" will be played each morning (daily) over the address system throughout the nursing home for approximately 5-10 minutes. Repeat CAPS tests will be obtained one week after the initiation of the study and at monthly intervals over a 12 month period of time. We propose to compare the posturographic data and the rate of falls recorded in the nursing homes to previously established fall data for the institutions. Preliminary observations have been associated with a decrease rate of falls in the geriatric nursing home environment when listening to the music of Nolwenn Leroy. The incorporation of these statistics will allow us to investigate a cost effective method of reducing falls that might save lives, evoke societal change and act as a model for other Geriatric Nursing Home settings. The objective measurements with the CAPS will allow us to further compare the incidence of falls with a probability of fall measurements.

ELIGIBILITY:
Inclusion Criteria:

* Geriatric Nursing Home Resident must be able to hear music

Exclusion Criteria:

* Deafness

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-02; Primary Completion 2006-04 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Dynamic Posturography | immediate pre and post music listening
Historical Falls related Institutional Data | From initial admissin to nursing home to present

CONTACTS AND LOCATIONS:
Overall Officials: Frederick R Carrick, PhD, FACCN, Study Director — Carrick Institute for Graduate Studies; Natalie J Engelbart, DC, DACNB, Principal Investigator — Carrick Institute for Graduate Studies; Michaele Sporaco, DC, Principal Investigator — Carrick Institute for Graduate Studies
Locations (1):
- Carrick Institute for Graduate Studies, Flower Mound, Texas, United States

IPD SHARING:
Plan to Share IPD: No